CLINICAL TRIAL: NCT01377051
Title: Acute Effect of Indacaterol Maleate on Static and Dynamic Lung Volume in COPD Subjects.
Brief Title: Effect of Indacaterol Maleate in Chronic Obstructive Pulmonary Disease (COPD) on Lung Volume and Related Dyspnea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Milan (Other)
Collaborators: Fondazione Salvatore Maugeri (Other)
Responsible Party: Principal Investigator, Pierachille Santus, MD, PhD, University of Milan
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 654CEC
Record Dates: First submitted 2011-06-15; First posted 2011-06-20 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: COPD; Lung Diseases; Dyspnea; Hypoxemia; Tachycardia
Keywords: COPD; Inspiratory capacity; Residual volume; Total lung resistance; Arterial Oxygen
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases; Dyspnea; Hypoxia; Tachycardia | interventions — indacaterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bronchodilator (Active Comparator): Indacaterol maleate 300 mcg will be administered by a third independent investigator following a randomization list.
  Interventions: Drug: Indacaterol maleate
- Placebo (Placebo Comparator): Will be administered with the same device by a third independent investigator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Indacaterol maleate — Dry powered, 300 mcg, only one inhalation with 24 hours duration
  Other Names: Onbrez, Hirobriz, Onbrize, Oslif Breezehaler, Arcapta
  Arms: Bronchodilator
Drug: Placebo — Dry powered, same to study drug, only one inhalation
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether indacaterol maleate 300 micrograms (mcg) is effective in the acute treatment of COPD and in particular on reducing lung hyperinflation and dynamic volumes.

DETAILED DESCRIPTION:
Enrolled patients: COPD of any disease severity in stable conditions. 48 hours of inhalatory drugs wash out.

Evaluation: Plethysmographic test, blood gas analysis, blood pressure, cardiac frequency and Borg scale evaluation in basal condition and after 60 minutes of indacaterol maleate 300 mcg inhalation.

ELIGIBILITY:
Inclusion Criteria:

* Signature of consensus
* COPD diagnosis
* Age from 50 to 85 years old
* history of COPD at least of one year
* respiratory stable conditions at least of one month
* Any basal FEV1 expressed in % of predicted value
* FEV1/ Forced Vital Capacity (FVC) less than 70%
* Former or active smokers with at least a smoking history of 20 pack year

Exclusion Criteria:

* Pregnancy
* FEV1/FVC more than 70%
* Known deficit of alpha 1 antitrypsin
* Subjects submitted to a Lung Volume Reduction Surgery (LVRS)
* Subjects with known positivity to Human Immunodeficiency Virus (HIV)
* Misuse of alcool or drugs
* Absence of compliance in performing respiratory tests

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-05; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Intra Thoracic Gas Volume (ITGV) | 60 minutes after drug inhalation
  A complete body plethysmografic test will be performed after indacaterol inhalation

SECONDARY OUTCOMES:
Forced Expired Volume in the first second (FEV1) | 60 minutes after drug inhalation
  Will be performed: spirometry, Arterial blood sample, measurement of blood pressure and cardiac frequency. All these parameters will be tested 60 minutes after inhalation of Indacaterol 300 micrograms (mcg).
Partial pressure of arterial oxygen (PaO2) | 60 minutes after drug inhalation
  Arterial gas analysis will be performed evaluating all arterial gases

CONTACTS AND LOCATIONS:
Overall Officials: Pierachille Santus, MD, PhD, Study Director — Università degli Studi di Milano-Pneumologia Riabilitativa- Fondazione Maugeri-Istituto Scientifico di Milano-IRCCS - pierachille.santus@unimi.it
Locations (1):
- Pneumologia Riabilitativa - Fondazione Maugeri - Istituto Scientifico di Milano - IRCCS, Milan, Italy